CLINICAL TRIAL: NCT00669773
Title: Phase 2 Randomized Study of Adriamycin & Docetaxel in the First-line Treatment of Locally Advanced or Metastatic Breast Cancer Patients With Measurable Primary Breast Tumor to Validate Gene Expression & Proteomic Signatures Predictive of Treatment Response
Brief Title: Validate Gene Expression and Proteomic Signatures Predictive of Treatment for Response for Breast Cancer Patient
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Haematology-Oncology, Dr. Lee Soo Chin, National University Hospital, Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BR08/34/06; HSA No: CTC0700019 (Other: Health Sciences Authority); 2006/00411 (Other: NHG Domain Specific Review Boards)
Record Dates: First submitted 2008-04-27; First posted 2008-04-30 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Docetaxel

ARMS (2):
- Adriamycin (Experimental): Arm A: 4 cycles of adriamycin at 75mg/m2 3 weekly followed by surgery followed by 4 cycles of docetaxel at 75mg/m2 3 weekly
  Interventions: Drug: Adriamycin
- Docetaxel (Experimental)
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Adriamycin — Arm A: 4 cycles of adriamycin at 75mg/m2 3 weekly followed by surgery followed by 4 cycles of docetaxel at 75mg/m2 3 weekly
  Arms: Adriamycin
Drug: Docetaxel — Arm B: 4 cycles of docetaxel at 75mg/m2 3 weekly followed by surgery followed by 4 cycles of adriamycin at 75mg/m2 3 weekly.
  Arms: Docetaxel

SUMMARY:
Primary Objectives

1. Validate our previously generated tumor gene expression and proteomic profiles in this independent sample to determine the predictive power to distinguish good from poor clinical and pathological responders to adriamycin or docetaxel.
2. Validate our previously generated plasma proteomic profiles in this independent sample to determine the predictive power to distinguish good from poor clinical and pathological responders to adriamycin and docetaxel.

Secondary objectives

1. To correlate adriamycin and docetaxel pharmacokinetics with

   1. Genetic polymorphisms of drug metabolizing enzymes and transporters, including MDR-1, Cyp3A, GSTs, and the nuclear receptors.
   2. Drug toxicity and tumor response.
   3. Peripheral mononuclear cell gene expression profiles
2. To study ondansetron pharmacokinetics and correlate that with genetic polymorphisms.

DETAILED DESCRIPTION:
Many chemotherapeutic agents are active in breast cancer, although response rate to any individual drug is only 30-50%. The choice of chemotherapy is empirical, and development of a chemosensitivity assay is desirable, to reduce costs, unnecessary toxicity, and loss of window of opportunity to cure. Single molecular markers to predict sensitivity are not highly accurate, as chemotherapy resistance mechanisms likely involve complex pathways. High-throughput technologies such as gene expression microarray and Proteinchip array allow simultaneous analysis of thousands of genes, and hundreds of proteins, and may be more informative. We previously conducted a study on patients with measurable primary breast tumor who received primary chemotherapy with an alternating regimen of adriamycin and docetaxel, and generated tumor genomic and tumor and plasma proteomic signatures that predicted for clinical and pathological response using high throughput discovery platforms. This protocol aims to recruit 20 patients as an independent test set to validate the genomic and proteomic signatures generated previously. Half the patients will be randomized to receive 4 cycles of pre-operative adriamycin (Arm A) allowing validation of the adriamycin-specific signatures, while the other half will be randomized to receive 4 cycles of pre-operative docetaxel (Arm B) allowing validation of the docetaxel-specific signatures. Subjects will then undergo resection of the primary breast tumor, followed by 4 cycles of adjuvant therapy with the alternative drug (docetaxel in Arm A, adriamycin in Arm B). Serial tumor and plasma samples will be obtained for genomic and proteomic analysis. The previously generated genomic and proteomic signatures will be applied to this independent dataset to categorize patients into good and poor responders, and the prediction correlated with actual treatment responses. Secondary goals include the correlation of patient genotype with drug pharmacokinetics, and the correlation of chemotherapy-induced peripheral blood mononuclear cell gene expression changes with treatment response and toxicities

ELIGIBILITY:
Inclusion Criteria:

Patients may be included in the study only if they meet all of the following criteria:

* Female, age 18 years or above.
* Histologic or cytologic diagnosis of breast carcinoma.
* T2-4 breast cancer with measurable primary breast tumor, defined as palpable tumor with both diameters 2.0cm or greater as measured by caliper.
* Patients must not have received prior chemotherapy or hormonal therapy for the treatment of breast cancer.
* Karnofsky performance status of 70 or higher.
* Estimated life expectancy of at least 12 weeks.
* Adequate organ function including the following:

  * Bone marrow:

    * Absolute neutrophil (segmented and bands) count (ANC)>= 1.5 x 10 9/L
    * Platelets >= 100 x 10 9/L
  * Hepatic:

    * Bilirubin <= 1.5 x upper limit of normal (ULN),
    * ALT or AST <= 2.5x ULN, (or <= 5 X with liver metastases)
  * Renal:

    * creatinine <= 1.5x ULN
* Left ventricular ejection fraction >= 50%
* Signed informed consent from patient or legal representative.
* Patients with reproductive potential must use an approved contraceptive method if appropriate (eg, intrauterine device, birth control pills, or barrier device) during and for three months after the study. Females with childbearing potential must have a negative serum pregnancy test within 7 days prior to study enrollment.

Exclusion Criteria:

Patients will be excluded from the study for any of the following reasons:

* Prior treatment for locally advanced or metastatic breast cancer.
* Treatment within the last 30 days with any investigational drug.
* Concurrent administration of any other tumor therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy.
* Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
* Pregnancy.
* Breast feeding.
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
* Poorly controlled diabetes mellitus.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* Symptomatic brain metastasis.
* History of significant neurological or mental disorder, including seizures or dementia.
* Peripheral neuropathy of CTC grade 2 or above (NCI CTC version 3).
* History of hypersensitivity to drugs formulated in Tween 80, the vehicle used for commercial docetaxel formulations.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-02; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Clinical and pathological response rate | 12 weeks
  Clinical and pathological response rate to four cycles of pre-operative chemotherapy.

SECONDARY OUTCOMES:
Baseline and serial changes in tumor & plasma genomic and proteomic changes | at different time-points (see description below)
  Core biopsy of breast tumor before treatment, after one cycle of pre-operative chemotherapy, and after the fourth cycle of pre-operative chemotherapy or study withdrawal for a total of 3 core biopsies.
  Plasma samples for proteomics before treatment, during pre-operative chemotherapy and before surgery, before first cycle of post-operative chemotherapy, within 4 weeks after completion of 4 cycles of post-operative chemotherapy, and four monthly thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Soo Chin LEE, MBBS, MRCP, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Chang JC, Wooten EC, Tsimelzon A, Hilsenbeck SG, Gutierrez MC, Tham YL, Kalidas M, Elledge R, Mohsin S, Osborne CK, Chamness GC, Allred DC, Lewis MT, Wong H, O'Connell P. Patterns of resistance and incomplete response to docetaxel by gene expression profiling in breast cancer patients. J Clin Oncol. 2005 Feb 20;23(6):1169-77. doi: 10.1200/JCO.2005.03.156. PMID 15718313
- [Background] Petricoin EF, Ardekani AM, Hitt BA, Levine PJ, Fusaro VA, Steinberg SM, Mills GB, Simone C, Fishman DA, Kohn EC, Liotta LA. Use of proteomic patterns in serum to identify ovarian cancer. Lancet. 2002 Feb 16;359(9306):572-7. doi: 10.1016/S0140-6736(02)07746-2. PMID 11867112
- [Derived] Voon PJ, Yap HL, Ma CY, Lu F, Wong AL, Sapari NS, Soong R, Soh TI, Goh BC, Lee HS, Lee SC. Correlation of aldo-ketoreductase (AKR) 1C3 genetic variant with doxorubicin pharmacodynamics in Asian breast cancer patients. Br J Clin Pharmacol. 2013 Jun;75(6):1497-505. doi: 10.1111/bcp.12021. PMID 23116553